CLINICAL TRIAL: NCT00247663
Title: Extension Study of 1.0mg Dose Letrozole Therapy in Postmenopausal Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345 1601
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Postmenopausal Women With Advanced Breast Cancer
Keywords: Aromatase inhibitor; letrozole; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Letrozole (Experimental)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole
  Other Names: FEM345

SUMMARY:
- To investigate the safety of letrozole monotherapy at a dose 1.0 mg/day or fadrozole monotherapy at a dose 2.0mg in Japanese postmenopausal patients with advanced breast cancer which participated in double blind study.

ELIGIBILITY:
Inclusion Criteria:

- Patients which participated in double blind study

Exclusion Criteria:

* Patients with intolerable toxicity.
* Patients which confirmed progressive disease during double blind study.
* Patients which have received concurrent anti-cancer therapy during double blind study.

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 1999-12; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Safety during treatment

SECONDARY OUTCOMES:
No secondary outcomes/objectives planned

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Japan (10):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Chuo-Ku, Tokyo
  - Novartis Investigative Site, Cyuo-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Nigata-honmachi
  - Novartis Investigative Site, Saitama